CLINICAL TRIAL: NCT03412422
Title: Ultrasound Assessment of Changes in the Diameter of the Common Carotid Artery After Increasing the Preload of the Heart With Passive Leg Raise and Intravenous Fluid Infusion
Brief Title: Ultrasound Assessment of Changes in the Diameter of the Common Carotid Artery After Increasing the Preload of the Heart
Status: Withdrawn | Type: Observational
Why Stopped: The study has been stopped due to technical difficulties.
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Maciej Piwoda, Principal Investigator, Uniwersytecki Szpital Kliniczny w Opolu
Other Study IDs: CCA_USG_PLR_USK
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Critical Illness; Fluid Responsiveness
Keywords: Passive Leg Raise; Fluid Challenge; Common carotid artery
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute circulatory failure: Mechanically ventilated patients with acute circulatory failure, monitored with PiCCO method, who need fluid responsiveness assessment.
  Interventions: Diagnostic Test: fluid responsiveness assessment

INTERVENTIONS:
Diagnostic Test: fluid responsiveness assessment — During the procedure, the investigator will be imaging one of the carotid arteries with ultrasound. In expiratory phase, four sets of three video loops will be recorded: before and after PLR and then before and after fluid challenge. There also will be noted hemodynamic parameters measured with PiCCO monitor. The fluid challenge is defined as administration of 500ml of crystalloid in less than 10 minutes. Later, another investigator, who will be blinded to other data, will measure the maximal and minimal diameter of CCA in each loop. The measurements will be averaged and eventually two values (maximal an minimal) from each set will be obtained.
  Other Names: passive leg raise; fluid challenge

SUMMARY:
Passive leg raise (PLR) and fluid challenge are useful tools in assessing the fluid responsiveness. However, they require continuous monitoring of cardiac output, which is usually an invasive technique and in some cases not always available. Vascular ultrasound can be an alternative to cardiac output monitoring in a fluid status evaluation. The common carotid artery (CCA) is an easily accessible vessel. It has recently been noted that the diameter of this artery changes after an intravenous fluid bolus. It is possible that the change in the diameter of the common carotid artery during passive leg raise and fluid challenge can be a predictor of fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated patients with circulatory failure, who are monitored with PiCCO and need fluid responsiveness assessment

Exclusion Criteria:

* contraindication for the volume administration (hydrostatic pulmonary edema or other evidence of fluid overload)
* contraindication for PLR test (e.g. after trauma)
* lack of possibility to examine the carotid arteries
* bilateral carotid surgery in the past
* bilateral anatomical defects of the carotid arteries
* unstable cardiac rhythm (e.g. atrial fibrillation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients admitted to critical care unit.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the diameter of the common carotid artery | 1 minute after PLR test and 1 minute after fluid challenge
  The diameter will be measured with ultrasound

SECONDARY OUTCOMES:
Evaluation the value of changes in the diameter of CCA as the predictor of fluid responsiveness. | 1 minute after PLR test and 1 minute after fluid challenge
  The changes in the diameter of CCA will be compared with the changes in cardiac output measured with PiCCO method.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu, Opole, Opole Voivodeship, Poland